CLINICAL TRIAL: NCT05930184
Title: Comparison of Laparoscopic Guided Peri-wound Transversus Abdominis Plane Block With Bupivacaine Versus Local Wound Infiltration on Post-op Opioid Use in Laparoscopic Sleeve Gastrectomy, A Prospective Randomized Controlled Study
Brief Title: Laparoscopic Guided Peri-wound Transversus Abdominis Plane Block With Bupivacaine Versus Local Wound Infiltration on Post-op Opioid Use in Laparoscopic Sleeve Gastrectomy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thanatat panitphong, Primary investigator, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HE651586
Record Dates: First submitted 2023-06-24; First posted 2023-07-05 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Morbid Obesity; Laparoscopic Sleeve Gastrectomy; Transversus Abdominis Plane Block; Local Wound Infiltration; Bupivacine; Opioid Use
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Periwound-TAP block using 0.25%Bupivacain 20ml and local wound infiltration using 0.25%Bupivacain 20ml
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local wound infiltration (Active Comparator): 0.25% Bupivacaine 20ml was injected into the wound subcutaneous tissue after the laparoscopic port was removed
  Interventions: Procedure: Local wound infiltration
- peri-wound Transversus Abdominis Plane Block (Experimental): 0.25% Bupivacaine 20ml was injected into the transversus abdominis plane around the wound before the laparoscopic port was removed
  Interventions: Procedure: peri-wound Transversus Abdominis Plane Block

INTERVENTIONS:
Procedure: peri-wound Transversus Abdominis Plane Block — 0.25% bupivacaine 20ml was injected using no24 needle into a plane between internal oblique muscle and transversus abdominis muscle around every wound 2 cm. from wound opening. The procedure was confirmed by laparoscopic vision and the injection was done before removal of laparoscopic port.
  Other Names: TAP block
  Arms: peri-wound Transversus Abdominis Plane Block
Procedure: Local wound infiltration — 0.25% bupivacaine 20ml was injected using no24 needle into subcutaneous tissue after the abdominal sheet was sutured.
  Arms: local wound infiltration

SUMMARY:
The goal of this randomized controlled trial is to compare laparoscopic guided peri-wound Transversus Abdominis Plane Block and bupivacaine versus local wound infiltration effect on reducing post-op opioid use in Laparoscopic Sleeve gastrectomy. The main questions it aims to answer are:

• Can laparoscopic guided peri-wound Transversus Abdominis Plane Block reduced post operative morphine usage when comparing with local wound port site infiltration.

Participants will be randomize into 2 group

* peri-wound Transversus Abdominis Plane Block
* local wound port site infiltration

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing LSG at Sringarind hospital as indicated by Thai guideline

Exclusion Criteria:

* Allergic/contraindicated to bupivacaine, morphine, fentanyl, NSAIDs or Nefopam
* Unable to describe pain score Opioid addict
* denied consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative morphine use | 48hours after intervention

SECONDARY OUTCOMES:
Post op VAS pain score | 48hours after intervention
length of hospital stay | within admission
opioid side effect | within admission
PACU time | 1day after intervention
postop complication | 2weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Thanatat Panitphong, Doctor of Medicine, Principal Investigator — Khon Kaen University
Locations (1):
- Srinagarind hospital, Khon Kaen, Northeastern, Thailand

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).